CLINICAL TRIAL: NCT05267964
Title: Trapeziometacarpal Prosthesis vs. Resection-Interposition Arthroplasty A Randomized Controlled Trial
Brief Title: Trapeziometacarpal Prosthesis vs. Resection-Interposition Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26-543 ex 13/14
Record Dates: First submitted 2022-01-24; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Arthropathy of Hand

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients are radomized into two groups prior to the surgical intervention using the radomizing programm of the medical university of graz.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epping resection arthroplasty (Active Comparator): During the Epping resection-suspension arthroplasty the trapeziectomy is performed, the flexor carpi radialis tendon is divided into two parts and one of these is stripped and cut proximally. To prevent shortening of the first ray with following loss of strength, this tendon strip is pulled through a drill hole in the base of the 1st metacarpal from ulnar palmar to radial dorsal. The rest of the tendon strip is sutured to a roll replacing the os trapezium.
  Interventions: Procedure: Epping resection arthroplasty
- CMC I prosthesis group (Active Comparator): During implantation of the prosthesis the CMC joint is opened and 3 mm of the metacarpal base as well as osteophytes are resected. Following the release of the trapezium the first metacarpal and the trapezium are prepared for the prosthesis by broaching and drilling. After the test-implants have shown satisfying joint tension and anatomic conditions, the HA coated stem and cup are pressfit inserted in the appropriate size followed by the modular head.
  Interventions: Procedure: CMC I prosthesis

INTERVENTIONS:
Procedure: Epping resection arthroplasty — Follwing the described epping resection arthroplasty, The first ray was immobilized using an orthosis for four weeks postoperatively in both study groups followed by eight weeks of physical therapy.
  Arms: Epping resection arthroplasty
Procedure: CMC I prosthesis — Follwing the described CMC I prosthesis procedure, The first ray was immobilized using an orthosis for four weeks postoperatively in both study groups followed by eight weeks of physical therapy.
  Arms: CMC I prosthesis group

SUMMARY:
Rhizarthrosis is a frequently occurring pathology leading to severe limitations in daily life due to pain and loss of function. Good clinical results have been reported for some carpometacarpal (CMC) joint prosthesis designs, but high failure rates due to loosening and dislocation must be considered. The study aim was to investigate a new, double mobility CMC-prosthesis design with special focus on (1) the functional outcome and (2) patient quality of life (QOL)

DETAILED DESCRIPTION:
The Epping resection-suspension arthroplasty procedure was described in 1983 to address the proximal migration of the first ray while providing pain free grip strength without any implants. It has shown rather good functional outcome and pain relief. A reduction in thumb opposition strength of 27% compared to the contralateral side and intermittent pain in physical activity is reported, however. Further, studies comparing trapeziectomy and trapeziectomy with tendon interposition recommend trapeziectomy due to the simple technique and comparable outcome.

Endoprosthesis of the first carpometacarpal (CMC) joint represents a different treatment strategy aiming at an exact reconstruction of the joint geometry. Some studies report excellent functional outcome and pain relief. However, there are some prosthesis designs (cemented and uncemented) with high rates of loosening, luxation and poor subjective results. To address these issues, a prosthesis was designed combining a cylindric, double mobility cup and a hydroxyapatite covered stem and cup available in different sizes. The aim of this study was to compare this new prosthesis design to the Epping arthroplasty as the current standard in the investigator's institution regarding (1) the functional outcome with special focus on mobility and strength and (2) patient quality of life (QOL) and pain relief.

Note: The registration of this trial on Clinicaltrials.gov was carried out retrospectively after primary completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic rhizarthrosis grade 2 and 3 according to Eaton's classification,
* failed conservative treatment prior to surgery,
* written informed consent to the study.

Exclusion Criteria:

* scaphotrapezotrapezoidal (STT) arthrosis,
* former CMC joint surgery,
* patients under custodianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome- Thumb opposition | twelve months postoperative
  Measurement of thumb opposition (scale from 1 to 10) range according to Kapandji.
  A score of 0 indicates no opposition, a score of 10 indicates maximal opposition.
Functional outcome - Thumb retropulsion | twelve months postoperative
  Measurement of thumb retropulsion (scale from 1 to 3) range according to Kapandji
Functional outcome - maximal palmar abduction | twelve months postoperative
  measurement of the maximal palmar abduction using a goniometer.
Functional outcome - maximal radial abduction | twelve months postoperative
  measurement of the maximal radial abduction using a goniometer.
Functional outcome - tip-to-tip force | twelve months postoperative
  The tip-to-tip force (between thumb and index finger) was measured in Newton (N) using a handheld dynamometer (Cit Technics, Haren, Netherlands).

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared at reasonable request.